## **DET VIDENSKABSETISKE KOMITÉSYSTEM**

(S1)

## Informeret samtykke til deltagelse i et sundhedsvidenskabeligt forskningsprojekt.

Forskningsprojektets titel: EDFI-Kohorten: Et kohortestudie om udviklingen af afføringsinkontinens og endetarmens lukkemuskels funktion, hos personer opereret for endetarmskræft.

## Erklæring fra forsøgspersonen:

Jeg har fået skriftlig og mundtlig information og jeg ved nok om formål, metode, fordele og ulemper til at sige ja til at deltage.

Jeg ved, at det er <u>frivilligt at deltage</u>, og at jeg altid kan trække mit samtykke tilbage uden at miste mine nuværende eller fremtidige rettigheder til behandling.

Jeg giver samtykke til, at deltage i forskningsprojektet, og har fået en kopi af dette samtykkeark samt en kopi af den skriftlige information om projektet til eget brug.

| rorsøgspersonens navn: |
|---|
| Dato: Underskrift: |
| Ønsker du at blive informeret om forskningsprojektets resultat samt eventuelle konsekvenser for dig?: |
| Ja (sæt x) |
| Erklæring fra den, der afgiver information: |
| Jeg erklærer, at forsøgspersonen har modtaget mundtlig og skriftlig information om forsøget. |
| Efter min overbevisning er der givet tilstrækkelig information til, at der kan træffes beslutning om<br>deltagelse i forsøget. |
| Navnet på den, der har afgivet information: |
| Dato: Underskrift: |
| Projektidentifikation: (Fx komiteens Projekt-ID, EudraCT nr., versions nr./dato eller lign.) |
| SJ-773 |